CLINICAL TRIAL: NCT00004769
Title: Myotonic Dystrophy:Muscle Wasting and Altered Metabolism
Brief Title: Study of Muscle Wasting and Altered Metabolism in Patients With Myotonic Dystrophy
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Richard T Moxley, Professor Of Neurology, University of Rochester
Other Study IDs: 199/11770; URMC-583 (Other: University of Rochester); URMC-445 (Other: University of Rochester)
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2013-01-28 (Estimated); Status verified 2013-01

CONDITIONS: Myotonic Muscular Dystrophy
Keywords: Genetic diseases; Myotonic muscular dystrophy; Facioscapulohumeral muscular dystrophy; CMT; Rare disease
MeSH Terms: conditions — Myotonic Dystrophy; Genetic Diseases, Inborn; Muscular Dystrophy, Facioscapulohumeral; Rare Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Myotonic dystrophy: Subjects with myotonic dystrophy
- Healthy controls: Healthy subjects
- Disease controls 1: Subjects with FSHD
- Disease controls 2: Subjects with CMT

SUMMARY:
OBJECTIVES: I. Examine the interrelationships between muscle wasting (phenotype), the degree of myotonic dystrophy (DM) gene expression (genotype) in patients with DM.

II. Characterize the insulin resistance in these patients. III. Assess the glucose uptake in the leg and forearm tissues of these patients.

IV. Determine the stability of the DM gene lesion in muscles over a 5-10 year period.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Patients are placed on a meatless diet 3 days prior to study entry.

During the first 5-day hospital stay, patients receive an oral glucose tolerance test, an intravenous glucose tolerance test, and an intravenous infusion of insulin and glucose (dextrose) to determine the degree of insulin resistance. Patients also receive dual x-ray absorptiometry (DEXA) scan and total body potassium count to measure muscle mass. Patients undergo strength testing and physical fitness screening. A needle biopsy is performed to investigate the genetic alterations associated with this disease.

During the second 3-day hospital stay, patients receive an intravenous infusion of insulin, stable isotopic glucose, and stable isotopic glycerol.

During the third 3-day hospital stay, a catheter is placed in the femoral artery, femoral vein, and in each arm. Patients receive an infusion of stable isotopic glucose, stable isotopic phenylalanine, and insulin. Measurements of the balance of amino acids and glucose across the forearm and leg are completed. Green dye is infused to measure blood flow in the leg.

ELIGIBILITY:
Inclusion Criteria:

* Clinically mild or moderate myotonic dystrophy (DM), proximal myotonic myopathy (PROMM), facioscapulohumeral muscular dystrophy (FSH) or, Charcot-Marie-Tooth (CMT)
* Mild or moderate DM defined as: Mild muscle weakness in the limbs, modest facial weakness, and mild grip myotonia; Moderate muscle weakness in the limbs, typical DM facies, and prominent grip myotonia

Exclusion Criteria:

* Prior or concurrent therapy
* Obese
* Concurrent acute illness

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: National sample
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 1993-12; Primary Completion 2000-03 (Actual); Study Completion 2000-03 (Actual)

PRIMARY OUTCOMES:
Quantitative myometry (QMT) | Visit 1

CONTACTS AND LOCATIONS:
Overall Officials: Richard T. Moxley, III, Study Chair — University of Rochester